CLINICAL TRIAL: NCT06232512
Title: Multimodal Haptic Feedback for Plantar Sensory Substitution
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Querrey Simpson Institute for Bioelectronics (Unknown); Northwestern University (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00218277
Record Dates: First submitted 2023-12-21; First posted 2024-01-30 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hypoesthesia
Keywords: Plantar Sensation
MeSH Terms: conditions — Hypesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exploratory Arm (Experimental): Individuals will complete standardized balance and walking tasks with and without sensory substitution from the haptic device system.
  Interventions: Device: Haptic Device

INTERVENTIONS:
Device: Haptic Device — Provides sensory substitution by mapping pressure from the insole sensor onto a corresponding vibrating and heating patch to be worn where more sensation is present.

SUMMARY:
The study will explore the use of a haptic device for sensory substitution in individuals with a movement disorder that has caused loss of plantar sensation. The haptic device consists of two components. The first element is a flexible insole with embedded pressure-sensing elements that transmit the spatial patterns of applied foot pressure over time. The second element is a haptic receiver with embedded actuators that vibrate or heat up in proportion to the transmitted pressure patterns, thus substituting the patient's lost plantar sensation.

DETAILED DESCRIPTION:
OBJECTIVES:

1. Identify a systematic, methodical approach to determine whether different users of our haptic device can perceive and use vibrational and thermal feedback in order to correct their posture in real-time.
2. Evaluate whether a haptic device can be used to guide users to maintain a prescribed pattern of pressure on their feet during standing and walking.
3. Investigate whether a haptic device can improve outcomes on motor evaluation tasks.

ELIGIBILITY:
Inclusion Criteria:

* Able to ambulate 10 meters with or without assistance
* Able and willing to give written consent and comply with study procedures

Exclusion Criteria:

* Unable to give written consent or comply with study procedures
* Unable to perceive unsafe levels of heat in relevant areas
* Has a motor complete spinal cord injury
* Have transfemoral (above knee) amputation
* Any condition that would prevent the safe completion of study activities, as determined by the Principal Investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pressure data from the insoles | During the intervention
  The primary outcome is to use the pressure-sensitive insole to ensure that we can accurately record spatial and temporal pressure data from a wide variety of healthy and non-healthy individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided